CLINICAL TRIAL: NCT04126109
Title: Parental Reports Toward in Vitro Fertilization
Brief Title: Parental Attitudes in Invitro Fertilization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Other Study IDs: In vito fertilizaion
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionaire — A questionaire will be offered to every parents

SUMMARY:
The relationship between revelation of mode of conception and child behavior is not known

DETAILED DESCRIPTION:
start of assisted reproductive techniques over the past 25 years made many otherwise infertile couples to become parents to genetically related children.

ELIGIBILITY:
Inclusion Criteria:

* Parents who were enrolled in ICSI and pregnancy occurred

Exclusion Criteria:

* ICSI with no pregnancy

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who are enrolled in ICI and became pregnant
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
The number of women who got pregnant that will tell others by that | within one year
  The number of women who got pregnant that will tell others by that method

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Algazeerah, Giza, Egypt